CLINICAL TRIAL: NCT03786887
Title: The 90% Effective Dose of Nalbuphine in Mechanical Ventilated Patients in the ICU
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hua-Qing Shu (Other)
Responsible Party: Sponsor-Investigator, Hua-Qing Shu, Associate chief physician, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HShu
Record Dates: First submitted 2018-12-03; First posted 2018-12-26 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-11

CONDITIONS: Pain
Keywords: mechanical ventilation; nalbuphine
MeSH Terms: conditions — Pain | interventions — Nalbuphine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nalbuphine (Experimental)
  Interventions: Drug: Nalbuphine

INTERVENTIONS:
Drug: Nalbuphine — dosage of nalbuphine

SUMMARY:
The aim of this study is to determine the effective nalbuphine dose in 90% of intubated patients in the ICU, including the continuous infusion dose and a bolus dose during moving to the lateral decubitus position. Pain will assessed using a Behavioural Pain Scale (BPS) requiring a score of 3-4.

DETAILED DESCRIPTION:
The continuous nalbuphine infusion dose starts at 100ug/kg/h, if the BPS scores reaches 3-4, the continuous infusion dose would be decreased by 20 ug/kg/h for next patients. If not, increased by 20 ug/kg/h.

The nalbuphine bolus is injected 5 min before turning the patients and the dose (starting at 0) is increased by 0.05 mg/kg, prior to each subsequent turn to lateral decubitus until a BPS score of 3-4 is obtained.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical invasive ventilation
* Sedated only with nalbuphine

Exclusion Criteria:

* Pregnant or breast-feeding woman
* Age below 18 or over 80 years
* An indication for deep sedation (e.g.the initial stage of septic shock, acute brain injury or acute respiratory distress syndrome)
* Renal dialysis
* The inability to assess pain by the BPS scale (e.g. paralysis)
* BMI less than 18 or more than 35
* Preadmission use of opioid analgesic for chronic pain
* Severe hepatic failure
* State of consciousness with impossibility to use self-assessment scale; monoamine oxidase inhibitors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10-24 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Continuous pumping dose of nalbuphine | 2 days
  The effective continuous infusion dose of nalbuphine to obtain a satisfactory analgesia
Nalbuphine bolus dose | 3 days
  The effective dose of a nalbuphine bolus to obtain a satisfactory analgesia

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Critical Care Medicine, Union Hospital, Wuhan, Wuhan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaveron D, Silva S, Sanchez-Verlaan P, Conil JM, Sommet A, Geeraerts T, Genestal M, Minville V, Fourcade O. The 90% effective dose of a sufentanil bolus for the management of painful positioning in intubated patients in the ICU. Eur J Anaesthesiol. 2012 Jun;29(6):280-5. doi: 10.1097/EJA.0b013e328352234d. PMID 22388706